CLINICAL TRIAL: NCT04168047
Title: Are Sleeping Disorders Associated With Visceral Hypersensitivity in Irritable Bowel Syndrome Patients ?
Acronym: S3i
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/381/HP
Record Dates: First submitted 2019-11-15; First posted 2019-11-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: visceral hypersensitivity; Insomnia
MeSH Terms: conditions — Irritable Bowel Syndrome; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy volunteers (Other)
  Interventions: Procedure: Barostat procedure; Other: Anxiety and Depression Evaluation; Other: Assessment of sleep quality
- Patients with insomnia (Other)
  Interventions: Procedure: Barostat procedure; Other: Anxiety and Depression Evaluation; Other: Assessment of sleep quality
- Patients with irritable bowel syndrome (Other)
  Interventions: Procedure: Barostat procedure; Other: Anxiety and Depression Evaluation; Other: Assessment of sleep quality
- Patients with irritable bowel syndrome and insomnia (Experimental)
  Interventions: Procedure: Barostat procedure; Other: Anxiety and Depression Evaluation; Other: Assessment of sleep quality

INTERVENTIONS:
Procedure: Barostat procedure — Pressure threshold will be measured during the barostat procedure
Other: Anxiety and Depression Evaluation — Anxiety and Depression will be measured using HAD anxiety and depression scale
Other: Assessment of sleep quality — Sleep quality will be measured using Pittsburg sleep quality index

SUMMARY:
Visceral hypersensitivity is frequent in IBS population up to 60% and is correlated with severity and altered quality of life. Sleeping troubles are most frequent in IBS population. Insomnia is a frequent disorder with an important cost for healthcare. Insomnia could decrease pain threshold.

Visceral hypersensitivity was never measure in patients with insomnia. The hypothesis is IBS patients with insomnia probably have lower visceral pain threshold.

The objective is to assess pain threshold during a barostat procedure in in IBS patients with or without insomnia in comparison with healthy volunteers or patients with insomnia.

If the hypothesis are confirmed, insomnia should be look at in IBS patients and its treatments could improve visceral hypersensitivity and IBS symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers

   - Person aged over 18 years with no IBS and no Insomnia
2. Patients with insomnia

   - Patient aged over 18 years with no IBS and no Insomnia
3. Patients with IBS

   - Patient aged over 18 years with IBS
4. patients with insomnia and IBS - Patient aged over 18 years with IBS

Exclusion Criteria:

* Active chronic organic disease
* Endometriosis
* Opioids consumption
* Change in chronic treatment in the last 30 days
* Hypersensitivity to Normacol
* Patient with blood dyscrasia disorder known or identified, anticoagulant or antiplatelet treatments
* Rectal pathology
* Intestinal occlusion
* Severe renal failure
* Sodium retention
* Anal pathology (anal fissure, hemorrhoidal thrombosis)
* Person with administrative or judicial decision or under legal protection measure
* Patient participating in another trial in the last 30 days
* Pregnant or breastfeeding women
* Impossibility to keep fasting for 12 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2025-11-12 (Actual); Study Completion 2025-11-12 (Actual)

PRIMARY OUTCOMES:
Pressure threshold measured during the barostat procedure | Day 35
  Pressure threshold measured during the barostat procedure

SECONDARY OUTCOMES:
Score at HAD anxiety and depression scale | Day 35
  Score at HAD anxiety and depression scale
Score at Pittsburg sleep quality index | Day 35
  Score at Pittsburg sleep quality index

CONTACTS AND LOCATIONS:
Overall Officials: Chloé MECHIOR, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No